CLINICAL TRIAL: NCT03545750
Title: Renal Replacement Anticoagulant Management
Acronym: RRAM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: University of Oxford (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Royal Surrey County Hospital NHS Foundation Trust (Other); University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: ICNARC/02/08/17
Record Dates: First submitted 2018-04-04; First posted 2018-06-04 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Critical Illness
Keywords: Acute kidney injury; Continuous renal replacement therapy; Citrate; Heparin
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regional citrate anticoagulation (RCA): Those receiving regional citrate anticoagulation for CRRT
- Systemic heparin anticoagulation (SHA): Those receiving systemic heparin anticoagulation for CRRT

SUMMARY:
Observational comparative effectiveness study of individual patient data using interrupted time series analysis techniques of linked data sources to establish clinical and health economic effects of moving from systemic heparin anticoagulation to regional citrate anticoagulation during continuous renal replacement therapy (CRRT) for patients treated on non-specialist Intensive Care Units (ICUs) in England and Wales.

DETAILED DESCRIPTION:
RRAM is an observational comparative effectiveness and cost-effectiveness study of individual patient data using interrupted time series analysis techniques and linked data sources. This study will use existing high quality clinical data collected for the Case Mix programme (CMP) - the national clinical audit for adult critical care - linked with Hospital Episodes Statistics, Office for National Statistics, and UK Renal Registry national data sets to establish the clinical and health economic effects of moving from systemic heparin anticoagulation (SHA) to regional citrate anticoagulation (RCA) during CRRT for patients treated on non-specialist ICUs in England and Wales. This will include data from approximately 85,000 patients treated with CRRT between 1 April 2009 and 31 March 2017 in 184 English non-specialist intensive care units within the ICNARC CMP.

Specific objectives of the RRAM are to:

1. Investigate the short-term benefits, risks, and costs of citrate anticoagulation.
2. Provide information on the subsequent development of end-stage renal disease (ESRD).
3. Trial the efficient research techniques, that if successful could be used to track the effects of any change in critical care practice occurring in ICUs in England and Wales over a reasonably short time scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or greater
* Admitted to an ICU participating in the ICNARC Case Mix Programme (CMP) in England between 1 April 2009 and 31st March 2017

Exclusion Criteria:

* Pre-existing end-stage renal disease (ESRD)
* Admitted to an ICU after kidney or kidney-pancreas transplantation
* Primary admission with acute hepatic failure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill adults who received CRRT on one or more day whilst treated on an ICU
Sampling Method: Non-Probability Sample
Enrollment: 85000 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 90-days
  All-cause mortality 90 days after first ICU admission in which CRRT was received
Incremental net monetary benefit | 1-year
  Incremental net monetary benefit gained at one year

SECONDARY OUTCOMES:
All-cause mortality | 30-days, and 1-year after ICU admission
  All-cause mortality at hospital discharge, 30 days and one year after ICU admission
Days of renal, cardiovascular, and advanced respiratory support whilst in ICU | Up to 5 years
  Total number of days receiving renal, cardiovascular, and advanced respiratory support
Bleeding and thromboembolic episodes | During index admission
  Occurrence of bleeding and thromboembolic episodes
ICU and hospital length of stay | Up to 5 years
  Length of stay in hospital and ICU
Dialysis-dependent renal disease | 1-year
  Identification of new dialysis-dependent renal disease at 1-year assessed by data linkage with UK Renal Registry
Estimated lifetime incremental net benefit associated with a change from heparin to citrate anticoagulation during CRRT | at 5 years
  Lifetime Incremental net monetary benefit gained

CONTACTS AND LOCATIONS:
Overall Officials: Peter Watkinson, MD, Principal Investigator — University of Oxford
Locations (1):
- Intensive Care National Audit and Research Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised study dataset will be availablefrom ICNARC on request to the Chief Investigator, subject to any necessary approvals

REFERENCES:
- [Derived] Gould DW, Doidge J, Zia Sadique M, Borthwick M, Caskey FJ, Forni L, Lawrence RF, MacEwen C, Mouncey PR, Ostermann M, Harrison DA, Rowan KM, Duncan Young J, Watkinson PJ. Renal replacement anticoagulant management: Protocol and analysis plan for an observational comparative effectiveness study of linked data sources. J Intensive Care Soc. 2022 Aug;23(3):311-317. doi: 10.1177/1751143720913417. Epub 2020 Apr 2. PMID 36033243
- [Derived] Gould DW, Doidge J, Sadique MZ, Borthwick M, Hatch R, Caskey FJ, Forni L, Lawrence RF, MacEwen C, Ostermann M, Mouncey PR, Harrison DA, Rowan KM, Young JD, Watkinson PJ. Heparin versus citrate anticoagulation for continuous renal replacement therapy in intensive care: the RRAM observational study. Health Technol Assess. 2022 Feb;26(13):1-58. doi: 10.3310/ZXHI9396. PMID 35212260